CLINICAL TRIAL: NCT07256379
Title: Clinical and Radiographic Evaluation of Implants in Protective Occlusion in Comparison to Normal Occlusion In Molars. A 2 -Years Randomized Clinical Trial.
Brief Title: Clinical and Radiographic Evaluation of Implants in Protective Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Dental Contiuing Education (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IDCE-16112025
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Implant Occlusion
Keywords: Implant Occlusion, protective occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protective occlusion (Active Comparator): According to the literature, Misch introduced the concept of implant-protective occlusion (IPO) (Misch and Bidez, 1994) based on basic prosthetic concepts, bone biomechanical principles and finite element analysis, which refers to an occlusal scheme designed for implant restoration, promoting the conditions for less biomechanical complications by reducing the stress to the implant interface and enhancing the longevity of the implant and prosthesis. It mainly entails the elimination of premature occlusal contacts or interferences.
  Interventions: Procedure: Protective occlusion
- Maximum Intercuspation (Experimental)
  Interventions: Procedure: Maximum Intercusption

INTERVENTIONS:
Procedure: Maximum Intercusption — to evaluate crestal bone loss, chewing efficiency and prosthetic complications after single posterior implant restoration in protective occlusion in comparison to maximum intercuspation occlusion.
  Arms: Maximum Intercuspation
Procedure: Protective occlusion — To evaluate crestal bone loss, chewing efficiency and prosthetic complications after single posterior implant restoration in protective occlusion in comparison to maximum intercuspation occlusion.
  Arms: Protective occlusion

SUMMARY:
Occlusal overload may lead to a number of complications; biological and mechanical such as crestal bone loss, screw loosening, prosthetic fracture and even implant failure . Inadequate occlusal scheme (occlusion) causes occlusal overload increasing mechanical stresses which are transferred to the crestal bone and implant interface, leading to complications such as; Early implant failure, Early crestal bone loss, Intermediate to late implant failure, Intermediate to late implant bone loss, Screw loosening (abutment and prosthesis coping), Uncemented restoration, Component fracture, Porcelain fracture, Prosthesis fracture and Peri implant disease .Thus, a proper implant occlusal scheme plays a major role in the outcome of the implant treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a single posterior (1st or second molar) bounded implant with opposing natural tooth teeth.
* Adults above the age of 18.
* Good oral hygiene.
* Patient accepts to provide informed consent.

Exclusion Criteria:

* Smokers.
* Pregnant and lactating females.
* Medically compromised patients.
* Patients with untreated active periodontal diseases.
* Patients with parafunctional habits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Loss | 2 years
  • To evaluate marginal bone loss using bitewing radiographs in mm.
Stability | 2 years
  • to assess implant micromotion in both groups by resonance frequency analysis (Osstell®) in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Continuing Education, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No